CLINICAL TRIAL: NCT02587715
Title: An Open-label, Non-randomized, Phase I/II Study of Allogeneic Human Umbilical Cord Tissue-Derived Mesenchymal Stem Cells (UC-MSC) and Liberation Therapy (When Associated With Chronic Cerebrovascular Venous Insufficiency) in Patients With Relapsing Remitting Multiple Sclerosis (RRMS)
Brief Title: A Study of Allogeneic Human UC-MSC and Liberation Therapy (When Associated With CCSVI) in Patients With RRMS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Novo Cellular Medicine Institute LLP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT/NOVO/2015/001
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AllogeneicHumanUmbilicalCordTissue-DerivedMesenchymalStemCells (Experimental): Super selective intravenous administration of 50 million Allogeneic Human Umbilical Cord Tissue-Derived Mesenchymal Stem Cells (UC-MSC) and intrathecal administration of UC-MSCs in dose of 100 million along with liberation therapy (when associated with CCSVI)
  Interventions: Biological: Allogeneic Human Umbilical Cord Tissue-Derived Mesenchymal Stem Cells; Other: Liberation therapy

INTERVENTIONS:
Biological: Allogeneic Human Umbilical Cord Tissue-Derived Mesenchymal Stem Cells — Super selective intravenous administration of 50 million Allogeneic Human Umbilical Cord Tissue-Derived Mesenchymal Stem Cells (UC-MSC) and intrathecal administration of UC-MSCs in dose of 100 million along with liberation therapy (when associated with CCSVI)
Other: Liberation therapy

SUMMARY:
STUDY OBJECTIVES:

Primary Objective: Assessment of treatment safety based on incidence of any treatment emergent/treatment associated adverse events prior to discharge and at 1, 3, 6 and 12 months post treatment.

Secondary objective: Assessment of efficacy at baseline, prior to discharge, 1 month, 3 months, 6 months and 12 months after treatment based on the following: EDSS and 29-item Multiple Sclerosis Impact Scale (MSIS-29), MS Functional Composite (MSFC) consisting of (1) Timed 25-Foot Walk, (2) 9 Hole Peg Test, and (3) Paced Auditory Serial Addition Test and gadolinium-enhanced magnetic resonance imaging (MRI)

DETAILED DESCRIPTION:
STUDY TREATMENT:

Investigational therapy product: Wharton Jelly derived allogeneic MSCs.

Method of administration and dose: Super selective intravenous administration of 50 million Allogeneic Human Umbilical Cord Tissue-Derived Mesenchymal Stem Cells (UC-MSC) and intrathecal administration of UC-MSCs in dose of 100 million along with liberation therapy (when associated with CCSVI).

SAFETY AND EFFICACY EVALUATION:

The proposed study will assess safety and primary and secondary efficacy endpoints after super selective intravenous and intrathecal administration of allogeneic umbilical cord mesenchymal stem cells (UC-MSC) in 69 patients with Relapsing Remitting Multiple Sclerosis.

Safety Evaluation:

Assessment of treatment safety based on incidence of any treatment emergent/treatment associated adverse events prior to discharge and at 1, 3, 6 and 12 months post treatment.

Efficacy evaluation:

Clinical evaluations, including EDSS and 29-item Multiple Sclerosis Impact Scale (MSIS-29) will be performed at baseline before stem cell mobilization, prior to discharge at 1, 3, 6 and 12 months after stem cell therapy.

The MS Functional Composite (MSFC) consists of the (a) Timed 25-Foot Walk, (b) 9 Hole Peg Test, and (c) Paced Auditory Serial Addition Test will be performed at baseline before stem cell mobilization and at 12 months after stem cell therapy.

Gadolinium enhanced MRI scans of the brain will be performed at baseline before therapy and then 12 months after stem cell therapy. Follow-up scans will be performed on the same type of scanner used at baseline. Scans will be analyzed centrally. The 'baseline MRI scan' will be the reference for brain volume changes.

DATA COLLECTION AND STATISTICAL ANALYSIS:

Descriptive analyses of the adverse events will be performed. Proportion of adverse events at each visit will be calculated using frequency distribution. The frequency, severity, timing and the potential relationship to the intervention will be assessed in order to characterize the safety of the intervention.

The probability of overall event-free survival (as well as progression-free, relapse-free, or MRI event-free survival) at baseline through 1 year will be calculated. The end point of progression is defined as increased Expanded Disability Status Scale (EDSS) score greater than 0.5 from baseline. Analyses will be conducted using Kaplan-Meier estimates with Wald-type 90% CIs based on Greenwood's formula for SE.

Descriptive analyses of all primary and secondary efficacy endpoints will be performed using descriptive statistics. Proportion of patients with clinically significant change in this efficacy measurement scales (EDSS, MSIS, MSFC, MSFC-25 foot walking test, MSFC-Nine Hole Peg Test, MSFC-Paced Auditory Serial Addition Test) and change in gadolinium enhancing lesions, new T2 lesions from previous visit will be presented as a proportion.

The percentage of change in brain volume will be calculated from screening and analyzed by end point status at month 12 with an exact Wilcoxon rank sum test using mean scores when the results are identical.The null hypothesis tests whether the median percentage of change in brain volume among participants who met the endpoint by month 12 is equal to the median of those who have not met the end point by month 12.

Other primary and secondary efficacy endpoints (EDSS, MSIS, MSFC, MSFC-25 foot walking test, MSFC-Nine Hole Peg Test, MSFC-Paced Auditory Serial Addition Test) will be analyzed using a Wilcoxon signed rank test. Change from baseline outcomes for all the endpoints will be calculated for each patient who underwent stem cell transplant as the post transplant value minus the baseline value. The null hypothesis tests whether the median difference from baseline measurement in the values at the month 1, month 3, month 6 and month 12 visits was significantly different from zero,with baseline measurement defined as the screening assessment for the percentage of change in brain volume and the baseline visit for all other end points.

To calculate MSFC, results from each of the 3 components will be transformed into a z score and averaged to yield a composite for each patient at each timepoint. The z scores that compose the MSFC score will be calculated using the reference population from the National Multiple Sclerosis Society Task Force database.

ELIGIBILITY:
Main inclusion criteria: Males and Females between age 18 and 60 years with confirmed diagnosis of Relapsing Remitting Multiple Sclerosis made by a neurology expert/MS expert with lesions demonstrated on brain MRI that are consistent with MS and having an EDSS (Kurtzke Expanded Disability Status Scale) score between 3.5 & 6

Inclusion Criteria:

* Males and Females between age 18 and 60 years
* Diagnosis of Relapsing Remitting Multiple Sclerosis made by a neurology expert/MS expert with lesions demonstrated on brain MRI that are consistent with MS
* Duration of disease: >5 years
* Having an EDSS (Kurtzke Expanded Disability Status Scale) score between 3.5 & 6
* History of 2 or more relapses within last 2 years with increase in EDSS scale of > 0.5 sustained for > 4 weeks
* Failure to respond or intolerance to the currently available Multiple Sclerosis (MS) immunomodulatory treatments): the lack of response to these treatments will be determined/defined by history of 2 or more relapses within last 2 years with increase in EDSS scale of > 0.5 sustained for > 4 weeks
* Must have proof of health insurance in country of residence

Exclusion Criteria:

* Primary progressive, secondary progressive or progressive relapsing MS as defined by Lublin and Reingold, 1996. These conditions require the presence of continuous clinical disease worsening over a period of at least 3 months. Subjects with these conditions may also have superimposed relapses but are distinguished from relapsing remitting subjects by the lack of clinically stable periods of clinical improvement.
* Unable to perform Timed 25-Foot Walk, 9 Hole Peg Test (HPT) (with both upper extremities) and Paced Auditory Serial Addition Test (PASAT 3)
* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease: For patients who have tested positive, an expert will be consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Patients with unstable cardiac status (unstable angina, attack of myocardial infarction within last 6 months, uncontrolled high blood pressure, hypotension, cardiomyopathy)
* Cerebrovascular accident within 6 months prior to study entry
* Patients with poorly controlled diabetes mellitus
* Patients with renal insufficiency (Creatinine> 2.5) or failure
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator is not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with clinical improvement in EDSS score compared to baseline | Up to 12 months
  Proportion of patients with clinical improvement in EDSS score compared to baseline.
  Clinical improvement is defined as decrease in Expanded Disability Status Scale (EDSS) score greater than 0.5 from baseline.

SECONDARY OUTCOMES:
Proportion of patients with a change in either gadolinium enhancing or new T2-weighted lesions on brain MRI | 12 months
Proportion of patients with reduction in T2 lesion volume on brain MRI | 12 months
Proportion of patients with reduction in brain volume on MRI | 12 months
Proportion of patients with clinical improvement in EDSS score compared to baseline | 3 months and 6 months
Proportion of patients with clinical improvement in MSIS score compared to baseline | 3 months, 6 months and 12 months
Proportion of patients with clinical improvement in MSFC score compared to baseline | 3 months, 6 months and 12 months
Proportion of patients with a change in mobility and leg function as measured by the 25 foot walking test | 12 months
Proportion of patients with a change in upper extremity function as measured by the Nine Hole Peg Test | 12 months
Proportion of patients with a change in cognitive function as measured by the Paced Auditory Serial Addition Test (PASAT) | 12 months
Proportion of patients with reduced number of relapses or freedom from progression of disease | 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Bill Brashier, M.D., Principal Investigator — Novo Cellular Medicine Institute LLP
Locations (1):
- Novo Cellular Medicine Institute, San Fernando, Trinidad, Trinidad and Tobago

REFERENCES:
- [Background] Bermel RA, Bakshi R. The measurement and clinical relevance of brain atrophy in multiple sclerosis. Lancet Neurol. 2006 Feb;5(2):158-70. doi: 10.1016/S1474-4422(06)70349-0. PMID 16426992
- [Background] Coles A. The curious incident of disability in multiple sclerosis trials. Lancet Neurol. 2006 Nov;5(11):899-900. doi: 10.1016/S1474-4422(06)70585-3. No abstract available. PMID 17052654
- [Background] Bjartmar C, Kidd G, Mork S, Rudick R, Trapp BD. Neurological disability correlates with spinal cord axonal loss and reduced N-acetyl aspartate in chronic multiple sclerosis patients. Ann Neurol. 2000 Dec;48(6):893-901. PMID 11117546
- [Background] Sormani MP, Arnold DL, De Stefano N. Treatment effect on brain atrophy correlates with treatment effect on disability in multiple sclerosis. Ann Neurol. 2014 Jan;75(1):43-9. doi: 10.1002/ana.24018. Epub 2014 Jan 2. PMID 24006277
- [Background] Till C, Ghassemi R, Aubert-Broche B, Kerbrat A, Collins DL, Narayanan S, Arnold DL, Desrocher M, Sled JG, Banwell BL. MRI correlates of cognitive impairment in childhood-onset multiple sclerosis. Neuropsychology. 2011 May;25(3):319-32. doi: 10.1037/a0022051. PMID 21534686
- [Background] Yaldizli O, Penner IK, Frontzek K, Naegelin Y, Amann M, Papadopoulou A, Sprenger T, Kuhle J, Calabrese P, Radu EW, Kappos L, Gass A. The relationship between total and regional corpus callosum atrophy, cognitive impairment and fatigue in multiple sclerosis patients. Mult Scler. 2014 Mar;20(3):356-64. doi: 10.1177/1352458513496880. Epub 2013 Aug 19. PMID 23959709
- [Background] Rudick RA, Lee JC, Nakamura K, Fisher E. Gray matter atrophy correlates with MS disability progression measured with MSFC but not EDSS. J Neurol Sci. 2009 Jul 15;282(1-2):106-11. doi: 10.1016/j.jns.2008.11.018. Epub 2008 Dec 19. PMID 19100997
- [Background] Barkhof F, Calabresi PA, Miller DH, Reingold SC. Imaging outcomes for neuroprotection and repair in multiple sclerosis trials. Nat Rev Neurol. 2009 May;5(5):256-66. doi: 10.1038/nrneurol.2009.41. PMID 19488083
- [Background] Popescu V, Agosta F, Hulst HE, Sluimer IC, Knol DL, Sormani MP, Enzinger C, Ropele S, Alonso J, Sastre-Garriga J, Rovira A, Montalban X, Bodini B, Ciccarelli O, Khaleeli Z, Chard DT, Matthews L, Palace J, Giorgio A, De Stefano N, Eisele P, Gass A, Polman CH, Uitdehaag BM, Messina MJ, Comi G, Filippi M, Barkhof F, Vrenken H; MAGNIMS Study Group. Brain atrophy and lesion load predict long term disability in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2013 Oct;84(10):1082-91. doi: 10.1136/jnnp-2012-304094. Epub 2013 Mar 23. PMID 23524331
- [Background] Pugliatti M, Rosati G, Carton H, Riise T, Drulovic J, Vecsei L, Milanov I. The epidemiology of multiple sclerosis in Europe. Eur J Neurol. 2006 Jul;13(7):700-22. doi: 10.1111/j.1468-1331.2006.01342.x. PMID 16834700
- [Background] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Background] Le Blanc K, Rasmusson I, Sundberg B, Gotherstrom C, Hassan M, Uzunel M, Ringden O. Treatment of severe acute graft-versus-host disease with third party haploidentical mesenchymal stem cells. Lancet. 2004 May 1;363(9419):1439-41. doi: 10.1016/S0140-6736(04)16104-7. PMID 15121408
- [Background] Kurtzke JF. Historical and clinical perspectives of the expanded disability status scale. Neuroepidemiology. 2008;31(1):1-9. doi: 10.1159/000136645. Epub 2008 Jun 6. PMID 18535394
- [Background] Rudick R, Antel J, Confavreux C, Cutter G, Ellison G, Fischer J, Lublin F, Miller A, Petkau J, Rao S, Reingold S, Syndulko K, Thompson A, Wallenberg J, Weinshenker B, Willoughby E. Recommendations from the National Multiple Sclerosis Society Clinical Outcomes Assessment Task Force. Ann Neurol. 1997 Sep;42(3):379-82. doi: 10.1002/ana.410420318. PMID 9307263
- [Background] Cutter GR, Baier ML, Rudick RA, Cookfair DL, Fischer JS, Petkau J, Syndulko K, Weinshenker BG, Antel JP, Confavreux C, Ellison GW, Lublin F, Miller AE, Rao SM, Reingold S, Thompson A, Willoughby E. Development of a multiple sclerosis functional composite as a clinical trial outcome measure. Brain. 1999 May;122 ( Pt 5):871-82. doi: 10.1093/brain/122.5.871. PMID 10355672
- [Background] Bonzano L, Roccatagliata L, Mancardi GL, Sormani MP. Gadolinium-enhancing or active T2 magnetic resonance imaging lesions in multiple sclerosis clinical trials? Mult Scler. 2009 Sep;15(9):1043-7. doi: 10.1177/1352458509106610. Epub 2009 Jul 1. PMID 19570818
- [Background] Kappos L, Moeri D, Radue EW, Schoetzau A, Schweikert K, Barkhof F, Miller D, Guttmann CR, Weiner HL, Gasperini C, Filippi M. Predictive value of gadolinium-enhanced magnetic resonance imaging for relapse rate and changes in disability or impairment in multiple sclerosis: a meta-analysis. Gadolinium MRI Meta-analysis Group. Lancet. 1999 Mar 20;353(9157):964-9. doi: 10.1016/s0140-6736(98)03053-0. PMID 10459905
- [Background] Brex PA, Ciccarelli O, O'Riordan JI, Sailer M, Thompson AJ, Miller DH. A longitudinal study of abnormalities on MRI and disability from multiple sclerosis. N Engl J Med. 2002 Jan 17;346(3):158-64. doi: 10.1056/NEJMoa011341. PMID 11796849
- [Background] O'Riordan JI, Gawne Cain M, Coles A, Wang L, Compston DA, Tofts P, Miller DH. T1 hypointense lesion load in secondary progressive multiple sclerosis: a comparison of pre versus post contrast loads and of manual versus semi automated threshold techniques for lesion segmentation. Mult Scler. 1998 Oct;4(5):408-12. doi: 10.1177/135245859800400502. PMID 9839300
- [Background] Chitnis T, Tardieu M, Amato MP, Banwell B, Bar-Or A, Ghezzi A, Kornberg A, Krupp LB, Pohl D, Rostasy K, Tenembaum S, Waubant E, Wassmer E. International Pediatric MS Study Group Clinical Trials Summit: meeting report. Neurology. 2013 Mar 19;80(12):1161-8. doi: 10.1212/WNL.0b013e318288694e. PMID 23509048
- [Background] Sormani MP, Bonzano L, Roccatagliata L, Cutter GR, Mancardi GL, Bruzzi P. Magnetic resonance imaging as a potential surrogate for relapses in multiple sclerosis: a meta-analytic approach. Ann Neurol. 2009 Mar;65(3):268-75. doi: 10.1002/ana.21606. PMID 19334061
- [Background] Sormani MP, Stubinski B, Cornelisse P, Rocak S, Li D, De Stefano N. Magnetic resonance active lesions as individual-level surrogate for relapses in multiple sclerosis. Mult Scler. 2011 May;17(5):541-9. doi: 10.1177/1352458510391837. Epub 2010 Dec 9. PMID 21148262
- [Background] Sormani MP, Bruzzi P, Beckmann K, Wagner K, Miller DH, Kappos L, Filippi M; European Study Group on Interferon Beta-1b in Secondary Progressive MS. MRI metrics as surrogate endpoints for EDSS progression in SPMS patients treated with IFN beta-1b. Neurology. 2003 May 13;60(9):1462-6. doi: 10.1212/01.wnl.0000063312.15758.b3. PMID 12743232
- [Background] Pascual AM, Martinez-Bisbal MC, Bosca I, Valero C, Coret F, Martinez-Granados B, Marti-Bonmati L, Mir A, Celda B, Casanova B. Axonal loss is progressive and partly dissociated from lesion load in early multiple sclerosis. Neurology. 2007 Jul 3;69(1):63-7. doi: 10.1212/01.wnl.0000265054.08610.12. PMID 17606882
- [Result] Klyushnenkova E, Mosca JD, Zernetkina V, Majumdar MK, Beggs KJ, Simonetti DW, Deans RJ, McIntosh KR. T cell responses to allogeneic human mesenchymal stem cells: immunogenicity, tolerance, and suppression. J Biomed Sci. 2005;12(1):47-57. doi: 10.1007/s11373-004-8183-7. PMID 15864738
- [Result] Le Blanc K, Tammik L, Sundberg B, Haynesworth SE, Ringden O. Mesenchymal stem cells inhibit and stimulate mixed lymphocyte cultures and mitogenic responses independently of the major histocompatibility complex. Scand J Immunol. 2003 Jan;57(1):11-20. doi: 10.1046/j.1365-3083.2003.01176.x. PMID 12542793
- [Result] Liu X, Zheng P, Wang X, Dai G, Cheng H, Zhang Z, Hua R, Niu X, Shi J, An Y. A preliminary evaluation of efficacy and safety of Wharton's jelly mesenchymal stem cell transplantation in patients with type 2 diabetes mellitus. Stem Cell Res Ther. 2014 Apr 23;5(2):57. doi: 10.1186/scrt446. PMID 24759263
- [Result] Watson N, Divers R, Kedar R, Mehindru A, Mehindru A, Borlongan MC, Borlongan CV. Discarded Wharton jelly of the human umbilical cord: a viable source for mesenchymal stromal cells. Cytotherapy. 2015 Jan;17(1):18-24. doi: 10.1016/j.jcyt.2014.08.009. Epub 2014 Oct 18. PMID 25442786
- [Result] Mikaeili Agah E, Parivar K, Joghataei MT. Therapeutic effect of transplanted human Wharton's jelly stem cell-derived oligodendrocyte progenitor cells (hWJ-MSC-derived OPCs) in an animal model of multiple sclerosis. Mol Neurobiol. 2014 Apr;49(2):625-32. doi: 10.1007/s12035-013-8543-2. Epub 2013 Aug 28. PMID 23982748